CLINICAL TRIAL: NCT07225712
Title: A Multicenter, Uncontrolled, Open-label Trial to Evaluate the Tolerability, Safety, and Efficacy of Long-term Administration of SEP-363856 in Patients With Schizophrenia
Brief Title: A Long-term Administration Trial of SEP-363856 in Patients With Schizophrenia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 382-102-00050
Record Dates: First submitted 2025-11-05; First posted 2025-11-10 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — SEP-363856

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- SEP-363856 75 or 100 mg/day (dose selected per protocol) (Experimental): SEP-363856 will be administered at 50 mg/day from Day 1 to Day 3, and 75 mg/day from Day 4 to Day 7. From Day 8 onward, the dose will, in principle, be 100 mg/day unless there are tolerability concerns; however, in accordance with protocol, the investigator or sub-investigator may select either 75 mg/day or 100 mg/day.
  Interventions: Drug: SEP-363856

INTERVENTIONS:
Drug: SEP-363856 — Tablet, once daily, for 52 weeks

SUMMARY:
To evaluate the safety of SEP-363856 (75 mg/day or 100 mg/day) administered for 52 weeks in adult participants with schizophrenia

ELIGIBILITY:
Inclusion Criteria:

* Japanese male or female participants 18 years of age or older at the time of informed consent
* Diagnosed with schizophrenia according to the DSM-5®
* Judged by the investigator to be clinically stable for at least 8 weeks prior to screening
* PANSS total score of 80 or less and CGI-S score 4 or less at both screening and baseline
* No changes in antipsychotic medication for at least 6 weeks before screening (excluding minor dose adjustments for tolerability)

Exclusion Criteria:

* History of psychiatric hospitalization within 8 weeks prior to screening
* Treatment-resistant to antipsychotic therapy (ie, within 1 year to screening, despite administration of two or more marketed antipsychotics at appropriate doses for at least 4 weeks [28 consecutive days] in accordance with the package insert, psychiatric symptoms did not improve)
* History of treatment with clozapine
* Unwillingness, before or during the trial period, to comply with the requirements for prior and concomitant medications/therapies as specified in the protocol or use of prohibited medications at screening or baseline as specified in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-22 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
・Incidence of treatment-emergent adverse events (TEAEs) | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nobuhito Sanada, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Jimbo Kokorono Clinic, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article Publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com.